CLINICAL TRIAL: NCT06550739
Title: Development and Validation of a New Prognostic System for Patients With Hepatocellular Carcinoma: A Cohort Study in China
Brief Title: Comprehensive Prognostic Model: The Study Introduces a Novel Prognostic Model That Incorporates a Wide Range of Clinical and Laboratory Variables, Providing a More Holistic Approach to Predicting Overall Survival in HCC Patients
Status: Completed | Type: Observational
Sponsor: Haike Lei (Other)
Responsible Party: Sponsor-Investigator, Haike Lei, Director, Chongqing University Cancer Hospital
Organization: Chongqing University Cancer Hospital (Other)
Other Study IDs: CZLS2023343-A
Record Dates: First submitted 2024-08-07; First posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Random Allocation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- training set: Patients were randomly divided into two groups: a training group of 671 individuals (approximately 70% of the data) and a validation group of 287 individuals (approximately 30% of the data).The nomogram model was developed using the training cohort.
  Interventions: Other: Randomization
- validation set: Validate the effectiveness of the model
  Interventions: Other: Randomization

INTERVENTIONS:
Other: Randomization — Randomly divide the data into a training set and a validation set in a 7:3 ratio

SUMMARY:
Background: Hepatocellular carcinoma (HCC) is a significant health problem in China, with high incidence and mortality rates. This study aimed to identify the prognostic factors of elderly HCC patients in southwest China and construct a new prognostic model for predicting overall survival (OS).

Methods: This retrospective cohort study collected clinical data from 958 patients with liver cancer on January 1, 2019, and December 12, 2020. The Cox regression model was used to test the significance of all available variables as prognostic factors of OS. Independent prognostic factors were identified based on multivariable analysis to model nomograms. The concordance index (C-index), the area under the receiver operating characteristic (AUC), the Time-dependent C-index, the Time-dependent AUC, the calibration curve, and decision curve analysis (DCA) were measured to assess the model performance of the nomogram.

Conclusions: The comprehensive risk prediction model for OS in HCC patients developed through this retrospective cohort study offers a promising avenue for improving clinical outcomes and patient care.

ELIGIBILITY:
Inclusion Criteria:

* (1) age ≥ 18 years; (2) had pathologically confirmed primary liver cancer; (3) received the main treatment in our hospital; (4) provided baseline clinical information and follow-up information; (5) completed the entire course of radiotherapy, chemotherapy and targeted therapy.

Exclusion Criteria:

* no follow-up records and a history of cancer treatments.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The data used in the retrospective cohort study were obtained from 958 patients with HCC from the Chongqing University Cancer Hospital tumor database between Jan 1, 2019, and Dec 12, 2020.
Sampling Method: Non-Probability Sample
Enrollment: 1053 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Survival status | April 31, 2024
  Patient survival or death

CONTACTS AND LOCATIONS:
Locations (1):
- Chongqing University Cancer Hospital, Chongqing, China

IPD SHARING:
Plan to Share IPD: No